CLINICAL TRIAL: NCT05507697
Title: Clinical Study of Human Umbilical Cord Mesenchymal Stem Cells in the Treatment of Refractory Diabetic Peripheral Neuropathy
Brief Title: Treatment With Human Umbilical Cord Mesenchymal Stem Cells for Refractory Diabetic Peripheral Neuropathy
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wuhan Central Hospital (Other)
Collaborators: Wuhan Optics Valley Vcanbio Cell & Gene Technology Co., Ltd., Hubei, China (Unknown); Wuhan Optics Valley Zhongyuan Pharmaceutical Co., Ltd., Hubei, China (Unknown)
Responsible Party: Principal Investigator, Shi Zhao, Principle Investigator, Clinical Professor, Wuhan Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WuhanCH
Record Dates: First submitted 2022-08-12; First posted 2022-08-19 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Diabetic Peripheral Neuropathy Type 2
Keywords: Diabetic Peripheral Neuropathy; Stem Cell; TCSS; Type 2 diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Thioctic Acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): MSCs Participants will received i. m. HUC-MSCs both lower extremities
  Interventions: Biological: HUC-MSCs
- Comparator (Placebo Comparator): The control group will receive i.v Lipoic Acid Injection
  Interventions: Biological: Lipoic Acid

INTERVENTIONS:
Biological: HUC-MSCs — 5 × 10^6 cells/mL, 1 mL per injection, each injection point is 2 cm apart ,1.0-1.5 cm deep, total amount of injection is estimated based on the surface area of the patient's lower limb
  Arms: Experimental
Biological: Lipoic Acid — Lipoic Acid Injection，600 mg/d for 15 consecutive days
  Arms: Comparator

SUMMARY:
Diabetic Peripheral Neuropathy (DPN) is one of the most common chronic complications in type 2 diabetes, conventional drug therapy can only target a single pathogenesis but not treat Diabetic Peripheral Neuropathy (DPN) fundamentally. As a novel technique, stem cell transplantation provides a new option for patients with DPN. In 2012, Wuhan Central Hospital, took the lead in carrying out clinical research on the treatment of DPN with autologous bone marrow stem cells in China, and patients were significantly relieved. Based on this research, our clinical trial is to evaluate the safety and efficacy of HUC-MSCs in the treatment of refractory diabetic peripheral neuropathy (DPN) by formulating standard operating procedures (SOP) and quality standards (QS) to explore the possible mechanism of HUC-MSCs in the treatment of DPN.

DETAILED DESCRIPTION:
As Diabetes is becoming a health problem of global concern rapidly, DPN, one of the common chronic complications in Diabetes is also getting more and more attention. The result of a survey of 5 regions in Southeast Asia showed that 39-72% of patients with DPN had severe or very severe impact on their quality of life. For the treatment of DPN, conventional drug therapy can almost only target a single pathogenesis and cannot treat it fundamentally. Therefore, new safe and effective treatment options for DPN are particularly important.

Both here and abroad, large number of experimental studies have shown that Bone Marrow or Umbilical Cord Mesenchymal Stem Cells have a significant therapeutic effect on diabetic peripheral neuropathy. In 2012, the Department of Endocrinology of Wuhan Central Hospital took the lead in conducting a clinical study of Autologous Bone Marrow Stem Cells in the treatment of DPN in China. The results of the study showed that the nerve conduction velocity of the lower extremities in most patients was improved within 3 months after treatment compared with before treatment. No serious adverse events occurred during the period. Based on this research of our own. The clinical trial is to evaluate the safety and efficacy of HUC-MSCs in the treatment of refractory diabetic peripheral neuropathy (DPN) by formulating standard operating procedures (SOP) and quality standards (QS) to explore the possible mechanism of HUC-MSCs in the treatment of DPN.

The investigators will do a Single center, randomization, open trial, controlled clinical trials design to assess treatment with the MSCs compared with the control group. 42 patients with DPN will be recruited in China. 21 patients receive i. m. HUC-MSCs both lower extremities (5 × 10^6 cells/mL, 1 mL per injection, each injection point is 2 cm apart ,1.0-1.5 cm deep, total amount of injection is estimated based on the surface area of the patient's lower limbs). 21 patients in the control group received i.v. Lipoic Acid Injection (600 mg/d for 15 consecutive days). Both efficacy and Adverse Event (AE) during the 96 weeks follow up.

ELIGIBILITY:
Inclusion Criteria:

* Ages at 18-55 years (including 18 and 55 years), regardless of gender;
* Understand and sign the ICF before proceeding with any steps related to this study, comply with the requirements, and do not to participate in other clinical studies during this research;
* T2DM patients defined by the 2013 American Diabetes Association (ADA) standards;
* Meet the diagnostic criteria for diabetic peripheral neuropathy: ① A clear history of diabetes; ② Neuropathy that occurs on or after the diagnosis of diabetes; ③Clinical symptoms and signs are consistent with DPN; ④ People with clinical symptoms (pain, numbness, abnormal sensation, etc.), had any 1 of the 5 items of ankle reflex, acupuncture pain, vibration, pressure and temperature in abnormal; people without clinical symptoms had any 2 of the 5 items were abnormal;
* The evaluation of symptoms and signs of neuropathy is at severe level (TCSS score ≥12);
* For conventional standard drug treatment (combined use of Lipoic Acid Capsules, Methyl cobalamin Tablets, and Epalrestat Tablets) at least 6 months and TCSS score decrease ≤30%;

Exclusion Criteria:

* Diseases that the investigator believes that it may interfere with subject compliance, including any uncontrolled diseases like in urinary, circulatory, respiratory, nervous, mental, digestive, endocrine, immune, and other system;
* Pregnant women, breastfeeding women or those who have a childbearing plan soon;
* Patients who are known to be allergic to cell products;
* People with various types of malignancies or hematological diseases;
* Complicated with severe lower extremity arterial disease (ankle-brachial index < 0.9)
* Complicated with foot ulcers, infections, or lower extremity amputation;
* Combined with neuropathy caused by other causes, such as lumbar spondylosis, cerebral infarction, Guillain-Barre Syndrome, excluding severe arteriovenous vascular disease, application of some chemotherapy drugs or renal insufficiency, etc. Nerve damage disease;
* Those who are unable or unwilling to provide informed consent or fail to comply with research requirements;
* Participated in other stem cell clinical researches before enrollment;
* Participated in other clinical trials within 3 months before enrollment.
* Patients with positive serum HIV antibodies;
* Patients with a history of alcohol and drug abuse and failed to abstain effectively

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2022-05-19 (Actual); Primary Completion 2024-05-18 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Change of TCSS scale | Change from Baseline TCSS scale at week 24
  1. Excellent: TCSS score decreased by >30% compared with the baseline value after treatment;
  2. Effective: TCSS score decreased by 30%-15% compared with the baseline value after treatment;
  3. Ineffective: Those who did not achieve the standards above after treatment.
Change of nerve conduction velocities in the lower extremity | Change from Baseline nerve conduction velocities in the lower extremity at week 12
  1. Excellent: after treatment, the lower extremity nerve conduction velocity and amplitude increased by more than 15% compared with the baseline value;
  2. Effective: after treatment, the lower extremity nerve conduction velocity and amplitude increased by 15%-5% compared with the baseline value;
  3. Ineffective: Those who did not achieve the standards above after treatment.

SECONDARY OUTCOMES:
Change of serum inflammatory factors | Baseline, week 4, week 12, week 24, week 36, week 48, week 96
  Observe the changes during the study period
Change of growth factors (GF) | Baseline, week 4, week 12, week 24, week 36, week 48, week 96
  Observe the changes during the study period
Change of fasting plasma glucose (FPG) | Baseline, week 12, week 24, week 36, week 48, week 96
  Observe the changes during the study period
Change of glycosylated hemoglobin (HbA1c) | Baseline, week 12, week 24, week 36, week 48, week 96
  Observe the changes during the study period

CONTACTS AND LOCATIONS:
Overall Officials: SHI ZHAO, Principal Investigator — Wuhan Central Hospital
Locations (1):
- The Central Hospital of Wuhan, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Yes
After approval from the steering committee and the Human Genetic Resources Administration of China, this trial data can be shared with qualifying researchers who submit a proposal with a valuable research question. A contract should be signed.